CLINICAL TRIAL: NCT00826618
Title: Pilot Study of Ranibizumab (Lucentis) for Uveitic Cystoid Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas Albini, Associate Professor of Clinical Ophthalmology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF4148s
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Uveitic Cystoid Macular Edema
Keywords: Uveitis; Cystoid Macular Edema
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — This is an open-label, Phase I study of intravitreally administered 0.5mg ranibizumab in subjects with uveitic CME.
  Other Names: Lucentis

SUMMARY:
Uveitic Cystoid Macular Edema (CME) is a major cause of visual loss associated with uveitis. Systemic and/or local corticosteroid therapy and systemic immunosuppression with steroid-sparing agents such as cyclosporine, methotrexate, azathioprine, or others, effectively treats uveitis and associated CME in many patients. However, in many cases, CME persists in spite of adequate suppression of uveitis. No consensus exists on how best to treat such cases. The further addition of immunosuppressive agents appears to have little effect on this form of CME. Oral corticosteroids are useful, but high dosage and prolonged use can be associated with serious side-effects. Periocular and intravitreal corticosteroid injections are associated with well-known, significant side effects such as glaucoma and cataract formation.

Vascular endothelial growth factor (VEGF) is suspected to play a role in the loss of vascular integrity in the eye and known to be induced by inflammatory cytokines, such as interleukin interleukin (IL)-1β and IL-6, which are elevated intraocularly in uveitis. In addition, it has been demonstrated that aqueous VEGF concentrations are statistically significantly higher in those uveitis patients with CME than those without CME. Inhibition of inappropriate VEGF activity is a potential approach to treatment of CME in uveitis given our current knowledge of the pathophysiology of this condition and also because of the clinical need for additional treatment options for these patients. Ranibizumab, a recombinant, humanized monoclonal antibody antigen-binding fragment (Fab) that neutralizes all active forms of VEGF-A, would target this pathway and may be useful in cases of persistent CME in uveitis patients.

The objective of this study is to determine if an anti-VEGF agent, Lucentis, is safe and effective in leading to regression of macular edema due to chronic non-infectious uveitis in patients with well-controlled uveitis.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

1. Ability to provide written informed consent and comply with study assessments for the full duration of the study.
2. Age > 18 years
3. Non-infectious uveitis in study eye.
4. Stable anti-uveitis medical regimen for at least one month prior to injection and controlled uveitis in the judgment of the investigator.
5. Vision 20/40 or worse in study eye.
6. Cystoid Macular Edema (CME) on fluorescein angiography (FA)
7. Optical Coherence Tomography (OCT) demonstrating thickness greater than 300 microns in the central subfield.
8. Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography.

Only one eye will be assessed in the study. If both eyes are eligible, the investigator will determine which eye will be entered into the study.

Exclusion Criteria:

1. Previous intravitreal triamcinolone injection in study eye within 3 months of study injection.
2. Use of more than two glaucoma medicines for study eye.
3. Significant epiretinal membrane as judged by treating physician.
4. Evidence of vitreomacular traction on OCT.
5. Previous vitrectomy in study eye.
6. Pregnancy (positive pregnancy test) or lactation.
7. Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an intrauterine device (IUD), or contraceptive hormone implant or patch.
8. Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
9. Participation in another simultaneous IND trial.
10. Treatment for CME with intravitreal Lucentis, Macugen, or Avastin within 6 weeks prior to enrollment in this study.
11. Uncontrolled inflammation in the study eye.
12. Current vitreous hemorrhage.
13. Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
14. Known allergy to any component of the study drug.
15. Intraocular pressure > 25 mm Hg despite treatment with glaucoma medications.
16. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, the subject can become eligible.
17. Major non-ocular surgery planned during the next 6 months.
18. Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
19. No Avastin use permitted in fellow eye during study.
20. Unwilling or unable to follow or comply with all study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Albini, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Bascom Palmer Eye Insitute, Miami, Florida
  - Bascom Palmer of the Palm Beaches, Palm Beach Gardens, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (19)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Early Treatment Diabetic Retinopathy Study (ETDRS at 4 Meters) at 12 Months.
Description: Mean change in best corrected visual acuity (assessed by the ETDRS chart at 4 m) from baseline at 12 months following first intravitreal injection of ranibizumab was 12.2 ETDRS letters (P = 0.015).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Change in ETDRS Letters
Groups:
- Ranibizumab: ranibizumab: This is an open-label, Phase I study of intravitreally administered 0.5mg ranibizumab in subjects with uveitic CME. Mean change in BCVA (assessed by the ETDRS chart at 4 m) from baseline at 12 months was 12.2 ETDRS letters (P = 0.015).
Arm/Group | Ranibizumab
Number analyzed (Participants) | 5
Change in ETDRS Letters | 12.2 (6.7)
Statistical Analysis 1: Comparison: Ranibizumab; Compare final visual acuity to baseline visual acuity; Test type: Superiority or Other; p = 0.0015, t-test, 2 sided

2. Secondary Outcome: The Mean Change in Best Corrected Visual Acuity (BCVA) (Assessed by the ETDRS Chart at 4 Meters) From Baseline at 12 Months Will be Computed With a T-test.
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: The Percentage of Patients With 15 Letters (3 Lines) of Visual Acuity Improvement at 30, 60, 90, 120 Days, and 12 Months.
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: The Mean Change in Foveal Retinal Thickness From Baseline at 7 Days, and at 30, 60, 90, 120 Days, and 12 Months Will be Computed Using a T-test.
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: The Incidence of Ocular and Non-ocular Adverse Events Will be Evaluated Through Month 24.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=5)
Floaters (Eye disorders) | 3
Eye Pain (Eye disorders) | 2
Blurry Vision (Eye disorders) | 2
Uveitis in fellow eye (Eye disorders) | 2
Anterior uveitis (Eye disorders) | 1
Dry Eye (Eye disorders) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Ocular pruritis (Eye disorders) | 1
Tachycardia (Cardiac disorders) | 1

LIMITATIONS AND CAVEATS:
The main limitation of this study is the small number of patients.There is no comparative arm to better define the relative efficacy of ranibizumab as compared with intraocular steroids or other treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No